CLINICAL TRIAL: NCT04662177
Title: Co-administration of Dexmedetomidine in Carotid Endarterectomy (CEA) With Intraoperative SSEP and MEP Monitoring: A Single-centre Prospective Randomized Controlled Trial
Brief Title: Co-administration of Dexmedetomidine in Carotid Endarterectomy (CEA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-00220
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomised controlled prospective trial in two groups. Group 1 will receive anaesthesia with propofol and co-administration of dexmedetomidine in conjunction with electrophysiological studies measuring somatosensory evoked potentials (SSEPs) and motor evoked potentials (MEPs). Group 2 will receive standard anaesthesia with propofol alone, in conjunction with electro¬physio¬logical studies measuring SSEPs and MEPs.
Who Masked: Participant
Masking Description: Randomised controlled prospective trial in two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Co-administration of dexmedetomidine and propofol with electrophysiological studies (Experimental): The group 1 starts with a bolus of dexmedetomidine 0.4 µg/kg over 10 minutes, followed by continuous infusion of dexmedetomidine 0.4 µg/kg/h until the end of burst suppression.
  Interventions: Drug: Dexmedetomidine
- Group 2: Standard anaesthesia with propofol and electrophysiological studies (No Intervention): The group 2 receive standard anaesthesia management.

INTERVENTIONS:
Drug: Dexmedetomidine — The study participants are divided into two groups: Group 1 starts with a bolus of dexmedetomidine 0.4 µg/kg over 10 minutes, followed by con-tinuous infusion of dexmedetomidine 0.4 µg/kg/h until the end of burst suppression. Group 2 receives the standard anaesthesia management.
  Other Names: Dexdor(R), Dexmedetomidine
  Arms: Group 1: Co-administration of dexmedetomidine and propofol with electrophysiological studies

SUMMARY:
All neurosurgical patients at the Neurosurgery University Hospital Bern who will be operated for carotid endarterectomy (CEA) are routinely operated in deep anae¬sthesia with suppression of the electrical activity of the electroencephalogram (EEG). To achieve this suppression of the EEG activity (burst suppression, BS) high effector concentrations (Cet) of Propofol doses are needed. However, a protracted infusion of large amounts of Propofol to reach a BS during the operation can lead to accumulation and a protracted wake-up phase with poorer neurological assessability. Somatosensory evoked potentials (SSEP), and trans-cranial Doppler flow velocity in the middle cerebral artery are measured to detect ischemia until the operation. The SSEPs are used to verify the functional integrity of the nervous system in combination of the EEG and both together exclude severe global ischemia during the operation.

The central acting α2-agonist Dexmedetomidine could help to reduce the amount of Propofol without influencing electrophysical studies. However, no data are currently known for practical use in carotid endarterectomy with Propofol with co-administration of Dexmedetomidine in conjunction with electrophysiological studies (SSEPs and MEPs).

DETAILED DESCRIPTION:
In the investigators clinic, as a neuroprotective measure, all neurosurgical patients operated for carotid endarterectomy (CEA) are routinely operated in deep anaesthesia with suppression of the electrical activity of the electroence-phalogram (EEG). To achieve this suppression of the EEG activity (burst suppression, BS) high effector concentrations (Cet) of Propofol doses are needed. However, a protracted infusion of large amounts of Propofol to reach a BS during the operation can lead to accumulation and a protracted wake-up phase with poorer neurological assessability.

Somatosensory evoked potentials (SSEP), and trans-cranial Doppler (TCD) flow velocity in the middle cerebral artery are measured to detect ischemia. A significant decrease in TCD velocity and/or SSEPs amplitudes during cross-clamping of the internal carotid artery (ICA) gets treated with an adapted increase of arterial blood pressure or placement of a shunt. Intraoperative monitoring and recording of data in every patient undergoing CEA median nerve SEPs and MCA flow velocity have been constantly monitored by an additional intraoperative monitoring (IOM) technician who has been trained and certified in the assessment of intraoperative monitoring. The median nerve SEP amplitudes are recorded at least at these events: baseline value before skin incision, EEG burst suppression before cross clamping of the internal carotid artery, at time of ICA cross clamping, 10 minutes after cross clamping or immediately after placement of shunt (ICA clamping), reperfusion of ICA and haemostasis / end of surgery. The predefined criterion for temporary shunting was the reduction of more than 50% of the SEP amplitude.

Median nerve somatosensory evoked potentials (SEPs) were performed by stimulation at the wrist with a pair of needle electrodes (Inomed Germany®). This is a single pulse stimulation with 0.5 ms pulse duration and a low repetition rate ranging from 0.7 - 2.3 Hz. Recording is performed via corkscrew electrodes placed accordingly to the 10-20-EEG system on the patient scalp. For the right median nerve SEP C3´/Fz and for the left median nerve SEP C4´/Fz is chosen as standard derivation. Alternatively, Cz' or the contralateral Cp' served as reference to improve quality of recording. To improve the signal to noise ratio the responses are averaged 150-200 times.

The investigator use the somatosensive evoked potentials (SSEPs) to verify the functional integrity of the nervous system. Standardized surgical and anaesthesiological measures at the CEA with defined EEG endpoints and depending on the anaesthetic effect can - in normal EEG and SSEPs - effectively exclude severe global ischemia. The effects of burst suppression and the volatile anaesthetics on SSEPs were also investigated and showed no significant difference. Since 2016, motor-induced evoked potentials (MEPs) have also been used, which are, however, suppressed by volatile anaesthetics in a dose-dependent manner. On the other hand, Dexmedetomidine in combination with Propofol seems to suppress only insignificantly.

The indication spectrum for the centrally acting α2-agonist Dexmedetomidine has been increasingly extended since its approval in Switzerland. In addition to the use of Dexmedetomidine in the intensive care units, Dexmedetomidine is also increasingly being used perioperatively up to premedication in children. In some studies, an anaesthetic reduction of 40-60% could be achieved or the opioid consumption after the addition of a α2-agonist could be reduced by 50-75%. The blood pressure response to a Dexmedetomidine dose depends on the rate of infusion). In addition, administration of Dexmedetomidine does not result in respiratory depression or compromising of the respiratory tract. It has been shown that Dexmedetomidine can cause a "sleep-like" sedation state and this state can be interrupted by verbal stimuli), examined the EEG activity in sedations on voluntary subjects compared to a control group with physiological sleep pattern. In this study, it was shown that the EEG spindle activity in subjects with Dexmedetomidine infusion was comparable to that of a physiological non-rapid eye-movement (nonREM) sleep stage II in the control tests. The authors concluded from their investigations that a "sleep-like state" (stage II non-REM) can be achieved by the Dexmed-etomidine infusion. However, no data are currently known for practical use in carotid endarterectomy with Propofol and Dexmedetomidine in conjunction with electrophysiological studies (somatosensory evoked potentials (SSEP) and motor evoked potentials (MEP)).

In addition, there is a high risk of postoperative delirium (POD) in many of these patients. This was examined in a recently published Lancet study by Xian Su and colleagues in 700 patients with non-cardiac interventions in elderly patients). A reduction of the delirium incidence from 23% to 9% was found after a low-dose Dexmedetomidine dose of 0.1 μg/kg body weight/h. In addition, Dexmedetomidine is attributed a neuroprotective effect against ischemic and hypoxic influences). Other animals-experimental studies indicate neuroprotection in ischemic insult and subsequent reperfusion).

ELIGIBILITY:
Inclusion criteria are:

* Age ≥18 years
* ASA physical status 1-4
* written informed consent provided.

Exclusion Criteria:

* Age <18 years
* higher grade atrioventricular block without pacemaker
* severe hypovolaemia or bradycardia
* uncontrolled hyper- or hypotension
* hypersensibility concerning the active substance dexmedetomidine or any other component
* serve liver disease
* known malignant hyperthermia
* cardiovascular instability or severe heart failure (> NYHA III)
* limited peripheral autonomic activity
* pregnancy
* rejection or lack of consent of the patient or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Effect size concentration of propofol. | until the operation
  The primary study outcome is to determine whether the intervention reduces the effect size concentration of propofol.

SECONDARY OUTCOMES:
intraoperative propofol requirement | until the operation
  the intraoperative propofol requirement or consumption, duration from end of surgery to extubation, intraoperative electrophysiological parameters , intraoperative haemodynamic parameters, vasoactive substances, and fluid management. We will also measure the vigilance, Richmond Agitation Sedation criteria for the development of delirium and muscle force of the extremities in the intensive care unit in the first 24 hours after the end of the operation at. Furthermore, we will examine the perioperative urinary output in these patients during the Operation. Additionally, we want to examine the patients' use of painkillers and the need for rescue analgesics as well as the postoperative nausea and vomiting direct after the patient has been extubated and once during the stay in the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Christian cv Vetter, MD, Principal Investigator — University of Bern
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetter C, Meyer ER, Seidel K, Bervini D, Huber M, Krejci V. Co-administration of dexmedetomidine with total intravenous anaesthesia in carotid endarterectomy reduces requirements for propofol and improves haemodynamic stability: A single-centre, prospective, randomised controlled trial. Eur J Anaesthesiol. 2025 Mar 1;42(3):255-264. doi: 10.1097/EJA.0000000000002099. Epub 2024 Nov 11. PMID 39529482

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT04662177/Prot_SAP_000.pdf